CLINICAL TRIAL: NCT05457725
Title: Characterizing and Modulating Neurocognitive Processes of Learning to Trust and Distrust in Aging II
Brief Title: Modulating Neurocognitive Processes of Learning to Trust and Distrust in Aging
Acronym: DecidingBrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202400337; R01AG072658 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Aging; Cognitive Change; Neurocognitive Disorders, Mild
Keywords: Decision Making; Trust; Learning; Socioemotional; Vulnerability to Exploitation
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Between subject design (experimental vs. control)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcome assessor are not aware of the experimental vs. control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contingent rtfMRI neurofeedback training (Experimental): Contingent rtfMRI neurofeedback training will follow an alternating up-regulation/rest block design with screen-color cues. Visual feedback about real-time brain activity in the ROI will be provided (e.g., via a thermometer bar). During resting blocks, the thermometer bar remains static.
  Interventions: Behavioral: Contingent rtfMRI neurofeedback training
- Non-contingent/sham rtfMRI neurofeedback training (Sham Comparator): Non-contingent/sham rtfMRI neurofeedback training will follow an alternating up-regulation/rest block design with screen-color cues. Visual feedback about non-contingent/sham brain activity in the ROI will be provided (e.g., via a thermometer bar). During resting blocks, the thermometer bar remains static.
  Interventions: Behavioral: Non-contingent/sham rtfMRI neurofeedback training

INTERVENTIONS:
Behavioral: Contingent rtfMRI neurofeedback training — Contingent rtfMRI neurofeedback training will follow an alternating up-regulation/rest block design with screen-color cues. Visual feedback about real-time brain activity in the ROI will be provided (e.g., via a thermometer bar). During resting blocks, the thermometer bar remains static.
  Arms: Contingent rtfMRI neurofeedback training
Behavioral: Non-contingent/sham rtfMRI neurofeedback training — Non-contingent/sham rtfMRI neurofeedback training will follow an alternating up-regulation/rest block design with screen-color cues. Visual feedback about non-contingent/sham brain activity in the ROI will be provided (e.g., via a thermometer bar). During resting blocks, the thermometer bar remains static.
  Arms: Non-contingent/sham rtfMRI neurofeedback training

SUMMARY:
Much of human interaction is based on trust. Aging has been associated with deficits in trust-related decision making, likely further exacerbated in age-associated neurodegenerative disease (Alzheimer's disease/AD), possibly underlying the dramatically growing public health problem of elder fraud. Optimal trust-related decision making and avoiding exploitation require the ability to learn about the trustworthiness of social partners across multiple interactions, but the role that learning plays in determining age deficits in trust decisions is currently unknown.

Aim: Probe the malleability of the underlying neurocircuitry of trust-learning deficits in aging. This study will utilize real-time fMRI neurofeedback to train older adults in brain activity up-regulation toward enhanced trust-related learning in aging and confirm critical mechanisms of experience-dependent social decisions in aging.

Grant R01AG072658 Aim 3: Test the malleability of trust-learning neurocircuitry toward optimized trust-related decision making in aging.

DETAILED DESCRIPTION:
This study will apply rtfMRI neurofeedback training as an intervention method, to demonstrate that older adults can be trained in volitional brain activity up-regulation, reducing their trust-learning deficits. The study will comprises several MRI sessions including pre-training, training, and post-training scans.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide verbal and written informed consent
* Fluent English speaker
* At least 8th grade education
* On stable medication regimen

Exclusion Criteria:

* Pregnancy
* Magnetic resonance imaging contraindications (e.g., certain metallic objects in body, claustrophobia)
* Current major depression defined as scores >14 on the Beck Depression Inventory-II
* Impaired scores on the Telephone Interview for Cognitive Status (TICS; cut-off of >30)
* Current use of medications with significant anticholinergic properties due to potential influence on memory ("memory enhancing"; e.g., Aricept or Namenda)
* Current use of anticonvulsant, neuroleptic, sedatives, or other medications known to affect cognition
* Uncorrected visual and hearing impairments
* Neurologic conditions affecting the brain (e.g., severe stroke, epilepsy, traumatic brain injury with >30-minute loss of consciousness)
* Impaired scores on a cognitive screening measure, the Montreal Cognitive Assessment (MoCA); for older adults the cutoff will be age and education corrected
* Unstable medical illness (e.g., metastatic cancer)
* Significant cardiovascular conditions (e.g., major heart attack)
* Will not exclude participants who are taking anti-depressant medications. Use of antidepressants (particularly SSRI's) and anxiolytic medications will be recorded and included in post-hoc analyses

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Neurofeedback Training Success | at baseline and after training completion about 1 week later
  Increase in BOLD signal in ROI during up-regulation trials administration of computerized learning tasks, with contrasting groups and conditions
Behavioral Benefits | at baseline and after training completion about 1 week later
  Increase in trust-related learning reflected in greater accuracy (e.g., in percent) on trust learning task

CONTACTS AND LOCATIONS:
Overall Officials: Natalie C. Ebner, PhD., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared with other researchers for secondary data analysis.